CLINICAL TRIAL: NCT05309213
Title: A Phase 1-2 Study to Evaluate the Safety and Efficacy of IM19 CAR-T Cells in Patients With Relapsed and Refractory (R/R) B-cell Acute Lymphoblastic Leukemia
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of IM19 CAR-T Cells in Patients With Relapsed and Refractory (R/R) B-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SD3
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Leukemia
Keywords: CAR-T; B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia; Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CAR-T cells (Experimental)
  Interventions: Biological: IM19 CAR-T cells

INTERVENTIONS:
Biological: IM19 CAR-T cells — IM19 CAR-T cells will be administered at dose level:5 x 10^4 CAR+ T cells/kg,1x 10^5 CAR+ T cells/kg,3 x 10^5 CAR+ T cells/kg,1 x 10^6 CAR+ T cells/kg

SUMMARY:
This is a phase I/II, open-label, multicenter study to assess the efficacy and safety of IM19 CAR-T cells in R/R B-cell Acute Lymphoblastic Leukemia

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-ALL, defined as:

  1. Not chieving a CR after 1 cycle of standard chemotherapy for relapsed leukemia.
  2. Any relapse after HSCT and must be ≥ 6 months from HSCT at the time of IM19 CAR-T cells infusion.
  3. Primary refractory as defined by not achieving a CR after 2 cycles of a standard chemotherapy regimen.
* Patients with Ph+ ALL are eligible if they are intolerant to or have failed two lines of TKI ± chemotherapy ；Ph + all patients with T315I mutation are not required to receive at least two TKI ± chemotherapy in the absence of effective TKI therapy;
* Morphological evidence of disease in bone marrow (at least 5% blasts).
* Aged 3 to 25 years, either sex;
* Estimated life expectancy >3 months;
* ECOG performance status of 0 or 1(age ≥ 16 years) or Lansky (age < 16 years) performance status ≥ 50;
* Women of childbearing age who had a negative blood pregnancy test before the start of the trial and agreed to take effective contraceptive measures during the trial period until the last follow-up; male subjects with fertility partners agreed to take effective contraceptive measures during the trial period until the last follow-up;
* Adequate organ function;
* Volunteer to participate in this trial and sign on the informed consent.

Exclusion Criteria:

* Isolated extramedullary disease relapse；
* Burkitt's lymphoma；
* Patient has obvious symptoms of central nervous system invasion and needs targeted treatment;
* Patient has previously received gene product therapy;
* Patients have graft-versus-host response（GVHD） and need to use immunosuppressants; Or GVHD ≥ grade 2 or being treated with anti GVHD; Or suffering from autoimmune diseases;
* Patient received chemotherapy or radiotherapy within 3 days before leukapheresis
* Patient used systemic steroids within 5 days before leucapheresis, except those who were recently or currently using inhaled steroids;
* Patients who used drugs to stimulate the production of bone marrow hematopoietic cells within 5 days before leucapheresis;
* Patients have participated in other clinical studies within 1 month before screening or plan to participate in other drug clinical trials during this study;
* Patient received allogeneic cell therapy within 6 weeks before CAR-T cell infusion, such as donor lymphocyte infusion(DLI)；
* History or presence of CNS disorder, such as epilepsy, epileptic seizures, cerebrovascular disease (ischemia / hemorrhage / cerebral infarction), brain edema, reversible posterior white matter encephalopathy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, cerebral organic syndrome or mental disease;
* Patients has HBV, HCV, HIV ,EBV,ECV or syphilis infection at the time of screening;
* Pregnant or lactating, or planning pregnancy within 180 days after the end of CAR-T cells infusion, or male patients whose partners plan pregnancy 180 days after their CAR-T cell infusion;
* Patients with other tumors in the past 5 years;
* Within 14 days before enrollment, there were active or uncontrollable infections requiring systemic treatment.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 28 days after CAR-T cell infusion
Persistence of CAR-T cells (cell counts and cell percentage in peripheral blood and bone marrow) | Up to 24 weeks after CAR-T cell infusion
  The persistence over time of CAR T cells in the peripheral blood as determined by flow cytometry and qPCR.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 28 days, 3 months and 6 months after CAR-T cell infusion
Anti-therapeutic IM19 CAR-T cells antibody | Up to 24 weeks after CAR-T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Qian Jiang, Principal Investigator — Peking University People's Hospital